CLINICAL TRIAL: NCT04369092
Title: Myotonometric Assessment of Muscles in Multiple Sclerosis Patients With Dysphagia
Brief Title: Myotonometer Analyses of Muscles in Multiple Sclerosis Patients With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuba Maden (Other)
Responsible Party: Sponsor-Investigator, Tuba Maden, Principal Investigator, clinical research, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/105
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis; Dysphagia; Swallowing Disorder; Deglutition Disorders; Muscle Tonus
MeSH Terms: conditions — Multiple Sclerosis; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- without swallowing problem (Other): patients without swallowing problem
  Interventions: Other: DYMUS
- mild swallowing problem (Other): patients with mild swallowing problem
  Interventions: Other: DYMUS
- severe swallowing problem (Other): patients with severe swallowing problem
  Interventions: Other: DYMUS

INTERVENTIONS:
Other: DYMUS — DYsphagia in MUltiple Sclerosis (DYMUS) that was questionnare and Eating Assessment Tool (EAT-10) were used for assess swallowing problem. All individuals were classified according to DYMUS. The DYMUS Score was 1 or 2 was taken as mild swallowing problems, 3 or more was taken as severe swallowing problems. Patients were divided into three groups; first group that include patients without swallowing problems, second group that include patients with mild swallowing problems, third group that include severe swallowing problems.
  Other Names: evaluating oropharyngeal dysphagia

SUMMARY:
Multiple Sclerosis is a chronic inflammatory autoimmune neurological disease characterized by the destruction of myelin in the central nervous system, grey matter and axonal loss. The prevalence of neurogenic dysphagia in this group of patients is estimated to be more than 30%. The aim of this study was investigating of Masseter, Orbicularis Oris, Sternocleidomastoid muscles' viscoelastic properties in MS patients with and without swallowing problems.

DETAILED DESCRIPTION:
The aim of this study was investigating of Masseter, Orbicularis Oris, Sternocleidomastoid muscles' viscoelastic properties in MS patients with and without swallowing problems. It carried out that myotonometric assessment of muscles in multiple sclerosis patients with dysphagia and comparison of these properties.

ELIGIBILITY:
Inclusion Criteria:

1. being diagnosed with Mc Donald's Multiple sclerosis (MS) in accordance with 2010 criteria,
2. being between the ages of 18-45.

Exclusion Criteria:

1. having psychological, orthopedic and other neurological disorders,
2. pregnancy,
3. having had an attack in the last 3 months,
4. application of botulinum toxin in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Myotonometric Measurement | through study completion, average one hour
  MyotonPro® device was used to measure muscles' viscoelastic parameters. The device is valid and reliable for measuring viscoelastic parameters (5, 6). Tonus, stiffness, elasticity of the muscles were recorded. Three measurements were bilaterally taken for each muscle. For each muscle, the average values of stiffness, tone and elasticity were retained as the main MyotonPRO outcomes. Myotonometric measurements were carried out for Masseter, Orbicularis Oris and Sternocleidomastoid (SKM) in supine position.

SECONDARY OUTCOMES:
Eating Assessment Tool | through study completion, average one hour
  Eating Assessment Tool was used to assess symptom of dysphagia. EAT-10 consisted of ten items, each of items was scored from 0 to 4. As the score increases, the patient's symptoms become deterioration.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)